CLINICAL TRIAL: NCT04022642
Title: Effects of a High-Intensity Interval Training Program Integrated in High-School Physical Education Classes, on Physical Condition, Physical Activity and Motivation for Exercise
Brief Title: Effects of HIIT Integrated in PE Classes, on Physical Condition, Physical Activity and Motivation for Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Principal Investigator, André Filipe Paulino da Silva Bento, Fellowship Researcher, University of Évora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SFRH/BD/136869/2018
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Adolescents
Keywords: HIIT; Adolescents; Physical Exercise; Health; Motivation
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Group (Experimental): Two HIIT sessions delivered at the beginning of Physical education classes
  Interventions: Other: High-Intensity Interval Training
- Control Group (No Intervention): Usual programmed Physical education classes

INTERVENTIONS:
Other: High-Intensity Interval Training — The program will be applied in the first 10-15 minutes of each PE class, twice a week, including a brief warm-up, ranged from 14 to 20 intervals, adopting a 2:1 work to rest ratio (ie, 30-s work, followed by 30-s rest)
  A cut-point of >=90% of maximal heart rate was used as our criterion for satisfactory compliance to high-intensity exercise
  In order to estimate effort, fatigue and training load, a subjective effort scale will be used throughout each session. The heart rate will be monitored throughout the session in real time through Bluetooth technology.
  Actigraph accelerometers (wGT3X-BT), randomly distributed by the students in each session, will be used to characterize the intensity of the sessions.
  Arms: HIIT Group

SUMMARY:
Levels of activity and physical condition among adolescents are low, increasing the risk of chronic diseases. The most recent literature suggests that physical activity and physical condition are correlated with improved biopsychosocial variables of the young. The School and, concretely, the Physical Education classes are privileged spaces, promoters of positive changes for the rest of the life. HIIT is an efficient alternative to the invested time compared to aerobic training, being a powerful stimulus in improving cardiorespiratory performance, muscles oxidative capacity and sensitivity to insulin. This study intends to verify the effectiveness and feasibility in the implementation of HIIT in High-School Physical Education classes. The activity levels and physical condition of the adolescents will be evaluated and identified, before and after 16 weeks of implementation of the training program, as well as their effects on the motivation for the practice.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in years 10-12

Exclusion Criteria:

* Students will be ineligible if they do not provide parental consent to participate

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline Cardio-respiratory fitness at 4 months | 4 months
  Assessed by Yo-Yo Intermitent Recovery Test 1(Tanner & Gore, 2014)
Change from 4 months Cardio-respiratory fitness at 6 months | 6 months
  Assessed by Yo-Yo Intermitent Recovery Test 1(Tanner & Gore, 2014)
Change from baseline Muscular Strength at 4 months | 4 months
  Assessed using push-up and curl-up tests (Plowman, 2013)
Change from 4 months Muscular Strength at 6 months | 6 months
  Assessed using push-up and curl-up tests (Plowman, 2013)
Change from baseline Body Mass Index (BMI) at 4 months | 4 months
  Assessed by Height and Weight (Dobbelsteyn, Joffres, MacLean, & Flowerdew, 2001)
Change from 4 months Body Mass Index (BMI) at 6 months | 6 months
  Assessed by Height and Weight (Dobbelsteyn, Joffres, MacLean, & Flowerdew, 2001)
Change from baseline Physical Activity at 4 months | 4 months
  Assessed by International Physical Activity Questionnaire (iPAQ), and accelerometry (Actigraph - wGT3X-BT)
Change from 4 months Physical Activity at 6 months | 6 months
  Assessed by International Physical Activity Questionnaire (iPAQ), and accelerometry (Actigraph - wGT3X-BT)
Change from baseline Motivation at 4 months | 4 months
  Assessed by Behavioral Regulation In Exercise Questionnaire (Cid et al., 2018).
Change from 4 months Motivation at 6 months | 6 months
  Assessed by Behavioral Regulation In Exercise Questionnaire (Cid et al., 2018).

CONTACTS AND LOCATIONS:
Overall Officials: André Bento, Principal Investigator — University of Évora
Locations (1):
- Escola Secundária D. Manuel I, Beja, Portugal